CLINICAL TRIAL: NCT01765543
Title: A Phase I, Open-Label, Multicenter, Three-Period, One-Sequence Study to Investigate the Effect of Rifampin on the Pharmacokinetics of a Single Oral Dose of 960 mg of Vemurafenib
Brief Title: A Pharmacokinetics (PK) Study to Investigate the Effect of Rifampin on PK of Vemurafenib (Zelboraf)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO28052; 2012-003142-33 (EudraCT Number)
Record Dates: First submitted 2013-01-09; First posted 2013-01-10 (Estimated); Results first posted 2016-12-15 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-10

CONDITIONS: Malignant Melanoma, Neoplasms
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — Rifampin; Vemurafenib

ARMS (1):
- Vemurafenib + Rifampin (Experimental): There will be 3 intervention periods in the study: Period A (Days 1 to 7), Period B (Days 8 to 16), and Period C (Days 17 to 24). Participants, after an overnight fast of at least 10 hours, will receive vemurafenib at a dose of 960 milligrams (mg) as film-coated tablets orally alone on Day 1 (Period A); with rifampin (at a dose of 600 mg as capsules orally) on Day 17 (Period C); and rifampin alone at a dose of 600 mg as capsules orally once daily will be administered from Days 8 through 16 (Period B) and from Days 18 through 23 (Period C).
  Interventions: Drug: Rifampin; Drug: Vemurafenib

INTERVENTIONS:
Drug: Rifampin — Rifampin at a dose of 600 mg as capsules orally once daily will be administered from Days 8 through 23 (Periods B and C).
Drug: Vemurafenib — Participants, after an overnight fast of at least 10 hours, will receive vemurafenib at a dose of 960 mg as film-coated tablets orally on Day 1 (Period A) and on Day 17 (Period C).
  Other Names: RO5185426, Zelboraf

SUMMARY:
This open-label, multi-center, three-period, one-sequence study will investigate the effect of rifampin on the PK of vemurafenib in participants with unresectable BRAFV600-mutation positive metastatic melanoma or other malignant tumor type that harbors a V600-activating mutation of BRAF without acceptable standard treatment options. Eligible participants will have the option to continue treatment with vemurafenib as part of an extension study GO28399 (NCT01739764).

ELIGIBILITY:
Inclusion Criteria:

* Participants with either unresectable Stage IIIc or Stage IV metastatic melanoma positive for the BRAF V600 mutation or other malignant tumor type that harbors a V600-activating mutation of BRAF, as determined by results of cobas® 4800 BRAF V600 mutation test or a Deoxyribonucleic acid (DNA) sequencing method, and who have no acceptable standard treatment options
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Life expectancy of greater than or equal to (>/=) 12 weeks
* Full recovery from the effects of any major surgery or significant traumatic injury within 14 days prior to the first dose of study treatment
* Adequate hematologic and end organ function
* Female participants of childbearing potential and male participants with partners of childbearing potential must agree to always use 2 effective methods of contraception
* Negative serum pregnancy test within 7 days prior to commencement of dosing in women of childbearing potential

Exclusion Criteria:

* Prior treatment with vemurafenib or other BRAF inhibitor within 42 days of first dose of study drug
* Requirement for immediate or urgent treatment with daily vemurafenib and for whom the intermittent schedule of vemurafenib employed during the 24-day period for this trial is not clinically acceptable
* Allergy or hypersensitivity to components of the vemurafenib formulation
* Experimental therapy within 4 weeks prior to first dose of study drug
* Major surgical procedure or significant traumatic injury within 14 days prior to first dose of study drug, or anticipation of the need for major surgery during study treatment
* Prior anti-cancer therapy within 28 days before the first dose of study drug
* History of clinically significant cardiac or pulmonary dysfunction
* History of symptomatic congestive heart failure of any New York Heart Association class or serious cardiac arrhythmia requiring treatment
* History of myocardial infarction within 6 months prior to first dose of study drug
* Current dyspnea at rest, owing to complications of advanced malignancy or any requirement for supplemental oxygen to perform activities of daily living
* History of congenital long QT syndrome or corrected QT interval (QTc) greater than (>) 450 milliseconds
* Active central nervous system lesions
* Uncontrolled or poorly controlled diabetes
* Current severe, uncontrolled systemic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- United States (4):
  - Rogers, Arkansas
  - Pleasant Hill, California
  - Middletown, Ohio
  - Dallas, Texas
- Porto Alegre, Rio Grande do Sul, Brazil
- Croatia (2):
  - Varaždin
  - Zagreb
- Egypt (4):
  - Alexandria
  - Cairo
  - Dakahlia
  - Tanta
- South Africa (2):
  - Cape Town
  - Port Elizabeth

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 27 participants were enrolled into the study.
Groups:
- Vemurafenib + Rifampin (All Periods): There were 3 intervention periods in the study: Period A (Days 1 to 7), Period B (Days 8 to 16), and Period C (Days 17 to 24). Participants, after an overnight fast of at least 10 hours, received vemurafenib (Zelboraf) at a dose of 960 milligrams (mg) as film-coated tablets orally alone on Day 1 (Period A); with rifampin (at a dose of 600 mg as capsules orally) on Day 17 (Period C); and rifampin alone at a dose of 600 mg as capsules orally once daily was administered from Days 8 through 16 (Period B) and from Days 18 through 23 (Period C).
Period: Overall Study
Arm/Group | Vemurafenib + Rifampin (All Periods)
Started | 27
Completed | 24
Not Completed | 3
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all participants who were enrolled in the study.
Groups:
- Vemurafenib + Rifampin (All Periods): There were 3 intervention periods in the study: Period A (Days 1 to 7), Period B (Days 8 to 16), and Period C (Days 17 to 24). Participants, after an overnight fast of at least 10 hours, received vemurafenib at a dose of 960 mg as film-coated tablets orally alone on Day 1 (Period A); with rifampin (at a dose of 600 mg as capsules orally) on Day 17 (Period C); and rifampin alone at a dose of 600 mg as capsules orally once daily was administered from Days 8 through 16 (Period B) and from Days 18 through 23 (Period C).
Arm/Group | Vemurafenib + Rifampin (All Periods)
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Time-curve From Zero to the Last Measurable Concentration Time Point (AUClast) of Vemurafenib
Description: AUClast is the area under the vemurafenib plasma concentration versus time curve from time zero to the time of last measured concentration of vemurafenib (Tlast). Area under the curve (AUC) is a measure of the plasma concentration of a drug over time. AUClast is presented in micrograms times (*) hour per milliliter (mcg*h/mL).
Time Frame: Predose (0 hour), 1, 2, 4, 6, 8, 12, 24, 30-32, 48, 72, 96, 120, 168 hours post vemurafenib-dose on Day 1 (Period A) and Day 17 (Period C)
Population: The pharmacokinetics (PK) parameter population included all participants who received both scheduled doses of vemurafenib and who provided adequate PK assessments to calculate important PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*h/mL
Groups:
- Vemurafenib (Intervention Period A): Participants, after an overnight fast of at least 10 hours, received vemurafenib alone at a dose of 960 mg as film-coated tablets orally on Day 1.
- Vemurafenib + Rifampin (Intervention Period C): Participants, after an overnight fast of at least 10 hours, received vemurafenib at a dose of 960 mg as film-coated tablets orally along with rifampin at a dose of 600 mg as capsules orally on Day 17 and rifampin alone at a dose of 600 mg as capsules orally once daily was administered from Days 18 through 23.
Arm/Group | Vemurafenib (Intervention Period A) | Vemurafenib + Rifampin (Intervention Period C)
Number analyzed (Participants) | 23 | 23
mcg*h/mL | 125 (101.4) | 76.7 (75.3)
Statistical Analysis 1: Comparison: Vemurafenib (Intervention Period A) vs Vemurafenib + Rifampin (Intervention Period C); Analysis of variance (ANOVA) was applied to the log-transformed PK parameters, and then back transformed to provide geometric mean ratio (Period C/Period A) and confidence intervals; Test type: Superiority or Other; Geometric Mean Ratio = 0.614, 90% CI 2-sided [0.484 to 0.780]

2. Primary Outcome: Area Under the Plasma Concentration Time-curve From Zero to Extrapolated Infinite Time (AUC[0-inf]) of Vemurafenib
Description: AUC(0-inf) is the AUC from time zero (pre-dose) to extrapolated infinite time (0-inf). AUC is a measure of the plasma concentration of a drug over time. AUC(0-inf) is presented in mcg*h/mL.
Time Frame: as for outcome 1
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*h/mL
Arm/Group | Vemurafenib (Intervention Period A) | Vemurafenib + Rifampin (Intervention Period C)
Number analyzed (Participants) | 23 | 23
mcg*h/mL | 131 (104.2) | 78.1 (74.3)
Statistical Analysis 1: Comparison: Vemurafenib (Intervention Period A) vs Vemurafenib + Rifampin (Intervention Period C); ANOVA was applied to the log-transformed PK parameters, and then back transformed to provide geometric mean ratio (Period C/Period A) and confidence intervals; Test type: Superiority or Other; Geometric Mean Ratio = 0.596, 90% CI 2-sided [0.469 to 0.759]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Vemurafenib
Description: Cmax is the maximum observed plasma vemurafenib concentration, presented in microgram per milliliter (mcg/mL).
Time Frame: as for outcome 1
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Vemurafenib (Intervention Period A) | Vemurafenib + Rifampin (Intervention Period C)
Number analyzed (Participants) | 23 | 23
mcg/mL | 4.45 (63.3) | 4.95 (59.1)
Statistical Analysis 1: Comparison: Vemurafenib (Intervention Period A) vs Vemurafenib + Rifampin (Intervention Period C); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Geometric Mean Ratio = 1.11, 90% CI 2-sided [0.908 to 1.36]

4. Other Pre Specified Outcome: Time to Reach Cmax (Tmax) of Vemurafenib
Description: Tmax is the time from vemurafenib administration to reach Cmax for vemurafenib.
Time Frame: as for outcome 1
Population: PK parameter population
Measure: Median (Full Range); unit: hours
Arm/Group | Vemurafenib (Intervention Period A) | Vemurafenib + Rifampin (Intervention Period C)
Number analyzed (Participants) | 23 | 23
hours | 4.00 [1.98 to 7.92] | 4.00 [1.98 to 6.02]

5. Other Pre Specified Outcome: Plasma Elimination Half Life (t1/2) of Vemurafenib
Description: Plasma elimination half-life is the time measured during drug elimination phase for the plasma drug concentration to decrease by one half.
Time Frame: as for outcome 1
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Vemurafenib (Intervention Period A) | Vemurafenib + Rifampin (Intervention Period C)
Number analyzed (Participants) | 23 | 23
hours | 29.7 (17.6) | 11.6 (5.24)

6. Other Pre Specified Outcome: Plasma Apparent Clearance (CL/F) of Vemurafenib
Description: Clearance of a drug is a measure of the rate at which a drug is removed (metabolized or eliminated by normal biological processes) from the blood. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Time Frame: as for outcome 1
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters/hour
Arm/Group | Vemurafenib (Intervention Period A) | Vemurafenib + Rifampin (Intervention Period C)
Number analyzed (Participants) | 23 | 23
liters/hour | 7.35 (104.2) | 12.3 (74.3)

7. Other Pre Specified Outcome: Area Under the Plasma Concentration Time-curve From Zero to 168 Hours [AUC(0-168)] of Vemurafenib
Description: AUC(0-168) is the AUC from time zero (pre-dose) to 168 hours (time point for last blood sample collection). AUC is a measure of the plasma concentration of a drug over time. AUC(0-168) is presented in mcg*h/mL.
Time Frame: as for outcome 1
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*h/mL
Arm/Group | Vemurafenib (Intervention Period A) | Vemurafenib + Rifampin (Intervention Period C)
Number analyzed (Participants) | 23 | 23
mcg*h/mL | 126 (99.6) | 78.0 (74.2)

8. Other Pre Specified Outcome: Percent Extrapolated AUC(0-inf) (AUCpeo) of Vemurafenib
Description: The AUCpeo, that is, percent area obtained after extrapolation from Tlast to infinity is calculated by using the formula AUCpeo = 100*(AUC[0-inf] minus AUC[0-last])/AUC(0-inf). This parameter provides information about what percentage of the theoretical curve AUC(0-inf) is possible to determine experimentally (AUC0-last).
Time Frame: as for outcome 1
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent AUC
Arm/Group | Vemurafenib (Intervention Period A) | Vemurafenib + Rifampin (Intervention Period C)
Number analyzed (Participants) | 23 | 23
percent AUC | 2.75 (150.4) | 1.26 (95.9)

ADVERSE EVENTS:
Time Frame: Day 1 up to 28 days after last dose of study drug (up to 51 days overall)
Description: The safety analysis population included all participants who received at least 1 dose of vemurafenib.
Groups:
- Rifampin (Intervention Period B): Participants received rifampin alone at a dose of 600 mg as capsules orally once daily from Days 8 through 16.
- Vemurafenib + Rifampin (Intervention Period C): Participants, after an overnight fast of at least 10 hours, received vemurafenib at a dose of 960 mg as film-coated tablets orally with rifampin at a dose of 600 mg as capsules orally on Day 17 and rifampin alone at a dose of 600 mg as capsules orally once daily was administered from Days 18 through 23.
Arm/Group | Vemurafenib (Intervention Period A) | Rifampin (Intervention Period B) | Vemurafenib + Rifampin (Intervention Period C) | Vemurafenib + Rifampin (All Periods)
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26 | 2/25 | 2/27
Other Adverse Events (participants affected / at risk) | 4/27 | 8/26 | 5/25 | 12/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib (Intervention Period A) (N=27) | Rifampin (Intervention Period B) (N=26) | Vemurafenib + Rifampin (Intervention Period C) (N=25) | Vemurafenib + Rifampin (All Periods) (N=27)
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib (Intervention Period A) (N=27) | Rifampin (Intervention Period B) (N=26) | Vemurafenib + Rifampin (Intervention Period C) (N=25) | Vemurafenib + Rifampin (All Periods) (N=27)
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2
Headache (Nervous system disorders) | 2 | 2 | 3 | 4
Chromaturia (Renal and urinary disorders) | 0 | 5 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.